CLINICAL TRIAL: NCT00889551
Title: Pregnancy and Growth of Adolescent Mothers and Their Child
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Brasilia (Other)
Other Study IDs: CEPFM 022/2003
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Adolescent; Pregnancy; Development

SUMMARY:
This study intends to observe the epidemiology of pregnancy and growth of adolescent mothers and their child in their first year on the development and growth ambulatory at Brasilia University Hospital (HUB).

The study hypothesis is that adolescent growth is disturbed by a pregnancy in this age. Another hypothesis is that their child's growth and development could be obstructed.

ELIGIBILITY:
Inclusion Criteria:

* in the HUB ambulatory of growth and development pediatric center

Exclusion Criteria:

* mothers who are more than 19 years old

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: adolescent mothers and their child that are in the ambulatory of growth and development in the pediatrics center of Braslia University Hospital - HUB
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Braslia University Hospital, Brasília, Federal District, Brazil